CLINICAL TRIAL: NCT02666027
Title: The Use of the Fluid IV Alert (FIVA) Monitor to Decrease the Incidence of Undetected Empty Intravenous Bag in Dimmed Operating Rooms
Brief Title: The Use of the Fluid IV Alert Monitor to Decrease the Incidence of Undetected Empty IV Bag in Dimmed Operating Rooms
Acronym: FIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Christian Lehmann, MD, PhD, FRCPC, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NSHA REB ROMEO File#: 1019905
Record Dates: First submitted 2015-11-05; First posted 2016-01-28 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia
Keywords: Fluid monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIVA ON (Experimental): The FIVA will be turned on for cases randomized to an even number. The ON light will be covered by tape. Routine induction and maintenance of anesthesia and rate and manner of delivery of IV fluid will be administered at the discretion by the anesthesiologist. The FIVA monitor will only monitor the first IV fluid bag since the study will be unblinded once the FIVA monitor alarm is triggered. When the IV bag is empty and the FIVA alarm is triggered, the anesthesiologist will turn off the FIVA and change the IV bag. The following will be recorded by the anesthesiologist: Type of surgical procedure; Duration of surgery; Presence of air in the IV; Number of false alarms triggered by the FIVA during the procedure; VAS assessment of ease of use of the FIVA; Loudness of audial alarm of the FIVA.
  Interventions: Device: Fluid Intravenous Alert (FIVA) 'on'
- FIVA OFF (Placebo Comparator): The FIVA will be off for cases randomized to odd numbers. The indicator lights will be covered by tape. Routine induction and maintenance of anesthesia and rate/manner of delivery of IV fluid will be administered at the discretion of the anesthesiologist. The IV bag may run dry with or without being noticed by the anesthesiologist. When they detect the empty bag, it will be changed after the removal of the FIVA. The anesthesiologist will record the presence or absence of air in the IV tubing following the termination of the study. The following will be recorded by the anesthesiologist: Type of surgery; Duration of surgery; Presence of air in the IV; Number of false alarms triggered by the FIVA device; VAS assessment of ease of use of the FIVA; Assessment of audial alarm of the FIVA.
  Interventions: Device: Fluid Intravenous Alert (FIVA) 'off'

INTERVENTIONS:
Device: Fluid Intravenous Alert (FIVA) 'on' — Fluid Intravenous Alert (FIVA) 'on' - The FIVA™ (EngenuityMED, Halifax, Canada) is a small, handheld, battery operated, device class I medical device in Canada (Figure 1). It is designed to alarm and alert the physician to change the IV bag when the fluid level in the chamber of the IV set is low. It also functions to stop the fluid flow through the gravity-fed tubing system when the alarm is triggered, preventing air from entering the IV tubing. We hypothesize that the FIVA would decrease the incidence of unnoticed dry IV bags during surgery, particularly when the operating room lights are dimmed and would therefore decrease the risks associated with undetected dry IV bags.
  Arms: FIVA ON
Device: Fluid Intravenous Alert (FIVA) 'off' — The FIVA will be turned off. - The FIVA™ (EngenuityMED, Halifax, Canada) is a small, handheld, battery operated, device class I medical device in Canada. It is designed to alarm and alert the physician to change the IV bag when the fluid level in the chamber of the IV set is low. It also functions to stop the fluid flow through the gravity-fed tubing system when the alarm is triggered, preventing air from entering the IV tubing. We hypothesize that the FIVA would decrease the incidence of unnoticed dry IV bags during surgery, particularly when the operating room lights are dimmed and would therefore decrease the risks associated with undetected dry IV bags.
  Arms: FIVA OFF

SUMMARY:
This study is being performed to determine the effectiveness of Fluid Intravenous Alert (FIVA) in monitoring intravenous fluid delivered to patients under anesthesia in a dimmed ambient light in the operating room.

DETAILED DESCRIPTION:
Background and Rationale

The first intravenous (IV) system was developed by Dr. Thomas Latta in 1832 to treat Cholera patients. Following its introduction, the IV delivery system has been widely adopted as a means of fluid resuscitation, rehydration and administration of blood products, medications and vasopressors. Today, it is a standard practice to place an IV catheter in all patients requiring an operation in the hospital setting. Intravenous fluid is administered through the IV tubing into the vein and carries the drugs that are needed for induction and maintenance of anesthesia. This IV fluid comes in several varieties which contain different amount of electrolytes, glucose, acidity or starch and is stored in a variety of volumes in sterile bags (most commonly 500 ml and 1000 ml). Once connected to the IV catheter through the IV tubing, the fluid bag is hung on the IV pole above the patient and flow into the patient by gravity.

In the nursing wards, IV fluids are routinely administered via infusion pumps, which can deliver fluid at specified rates and volumes and would sound alarms when the selected volumes of fluid have been completed. While this is an effective means of administering IV fluid, it is a time-consuming process to set up the IV fluid pump and program the infusion volume and rate. Perioperative fluid administration is a rapidly changing process and most anesthesiologists would prefer more control over the rate than pre-programed pumps. In the operating room environment, the rate and manner of drug and fluid administration are highly variable. Therefore, almost all IV fluid administered systems are gravity-fed.

In busy operating rooms, anesthesiologists carefully observe the progress of surgery and the anesthetic state of patients through different monitors. Intravenous fluid bags often run empty unnoticed because the IV fluid bags are hung above the eye level of the anesthesiologist. Even a vigilant anesthesiologist may not be able to promptly detect dry the IV fluid bag. In a previous observational study, the incidence of undetected dry IV bags has been shown to be 29.6%. However, the length of time before an empty bag is noticed is unknown. According to a recent survey about the working conditions in the operating room, including 471 surgeons and 405 nurses, most of the reported intra-operative hazards were due to insufficient illumination of the operating room especially during dangerous situations, such as unexpected bleeding. In the presence of dimmed ambient light in the operating room, e.g. during endoscopic surgeries, it is probably more difficult to visually monitor the flow of IV fluid with higher incidence of undetected dry IV bags. Several potential clinical adverse events can occur if the dry IV bag is not detected promptly. Firstly, if the gravity-fed IV fluid is being used as a carrier to administer drugs, such as anesthetics for total intravenous anesthesia (TIVA), or the infusion of vasopressors, awareness under anesthesia or unstable hemodynamics may occur. Secondly, during fluid or volume resuscitation, the IV fluid delivery system is frequently pressurized in order to deliver fluid as quickly as possible to the unstable patient. The pressurized IV fluid bag can force the air present in the IV fluid bag into the IV tubing when the fluid runs out. This can potentially cause air embolism. Finally, undetected dry IV bags can disrupt fluid flow through the catheter into the patient, allowing blood to pool around the catheter. If a clot is formed, it will occlude the line and prevent any further fluid flow. This may necessitate recannulation of the anesthetized patient during surgery which may be technically challenging.

The FIVA™ (EngenuityMED, Halifax, Canada) is a small, handheld, battery operated, device class I medical device in Canada. It is designed to alarm and alert the physician to change the IV bag when the fluid level in the chamber of the IV set is low. It also functions to stop the fluid flow through the gravity-fed tubing system when the alarm is triggered, preventing air from entering the IV tubing.

We hypothesize that the FIVA would decrease the incidence of unnoticed dry IV bags during surgery, particularly when the operating room lights are dimmed and would therefore decrease the risks associated with undetected dry IV bags.

ELIGIBILITY:
Inclusion Criteria:

- Attending anesthesiologists scheduled for elective surgical procedures at the Queen Elizabeth II Health Sciences Centre (QEII).

Exclusion Criteria:

* Attending anesthesiologists scheduled for elective surgical procedures at the QEII with cases where lights to not dimmed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence of undetected dry IV bags | For the duration of the surgery

SECONDARY OUTCOMES:
Type of surgical procedure | Baseline
  Questionnaire
Duration of surgical procedure | Baseline
  Questionnaire
Presence of air in the IV | For the duration of surgery
  Questionnaire
Number of false alarms triggered by the FIVA device during the procedure | For the duration of surgery
VAS assessment of ease of use of the FIVA | For the duration of surgery
Loudness of audial alarm of the FIVA | For the duration of surgery
  Questionnaire
Ease of use of the FIVA | For the duration of surgery
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christian Lehmann, MD, PhD, Principal Investigator — Nova Scotia Health Authority

REFERENCES:
- [Background] Janakan G, Ellis H. Dr Thomas Aitchison Latta (c1796-1833): pioneer of intravenous fluid replacement in the treatment of cholera. J Med Biogr. 2013 May;21(2):70-4. doi: 10.1258/jmb.2012.012004. PMID 24585745
- [Background] Matern U, Koneczny S. Safety, hazards and ergonomics in the operating room. Surg Endosc. 2007 Nov;21(11):1965-9. doi: 10.1007/s00464-007-9396-4. Epub 2007 May 5. PMID 17483989
- [Background] Hung OR, Comeau. L. Incidence of intra-operative cessation of intravenous (iv) fluid administration. Can J Anesth 1998;45:A5.
- [Background] Mendenhall ML, Spain DA. Venous air embolism and pressure infusion devices. J Trauma. 2007 Jul;63(1):246. doi: 10.1097/01.ta.0000210439.64958.df. No abstract available. PMID 17622901
- [Background] Mirski MA, Lele AV, Fitzsimmons L, Toung TJ. Diagnosis and treatment of vascular air embolism. Anesthesiology. 2007 Jan;106(1):164-77. doi: 10.1097/00000542-200701000-00026. PMID 17197859
- [Background] Pant D, Narani KK, Sood J. Significant air embolism: A possibility even with collapsible intravenous fluid containers when used with rapid infuser system. Indian J Anaesth. 2010 Jan;54(1):49-51. doi: 10.4103/0019-5049.60498. PMID 20532073